CLINICAL TRIAL: NCT06463808
Title: Effect of Recombinant Human Brain Natriuretic Peptide on Ventricular Remodeling and Cardiac Function in Patients With Acute Anterior Myocardial Infraction Undergoing Percutaneous Coronary Intervention
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: REBUILD-AAMI
Record Dates: First submitted 2023-12-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Ventricular Remodeling; Myocardial Infarction, Anterior Wall
Keywords: Myocardial Infarction, Anterior Wall; Recombinant Human Brain Natriuretic Peptide; Ventricular Remodeling; Percutaneous Coronary Intervention
MeSH Terms: conditions — Ventricular Remodeling; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who take Recombinant Human Brain Natriuretic Peptide
  Interventions: Drug: Recombinant Human Brain Natriuretic Peptide
- patients who do not take Recombinant Human Brain Natriuretic Peptide

INTERVENTIONS:
Drug: Recombinant Human Brain Natriuretic Peptide — we divide our subjects into two groups;one is required to take recombinant human brain natriuretic peptide,the other is not required to take recombinant human brain natriuretic peptide
  Groups: patients who take Recombinant Human Brain Natriuretic Peptide

SUMMARY:
This study is designed to evaluate the efficacy and safety of Recombinant Human Brain Natriuretic Peptide (rhBNP) in improving ventricular remodeling and cardiac function after acute anterior myocardial infarction undergoing percutaneous coronary intervention. 100 patients with acute anterior myocardial infarction after primary Percutaneous Coronary Intervention (pPCI) are randomly assigned 1:1 to rhBNP group(n=50) and control group(n=50) with follow-up of 24 weeks. Both groups are treated with standard therapy of AAMI, with the rhBNP group intravenous dripping rhBNP after pPCI for 3 days and the control group treated with placebo at the same time. The primary endpoint is the change in N terminal pro-B-type natriuretic peptide（NT-proBNP ）and cardiac troponin T(cTnT) level.The secondary endpoint is the change in 24-week echocardiographic including left ventricle ejection fraction (LVEF) , left ventricular end-diastolic volume index (LVEDVI) and left ventricular end-systolic volume index (LVESVI), arrhythmia and cardiovascular events (death, cardiac arrest or cardiopulmonary resuscitation, hospitalization due to heart failure or angina pectoris).

ELIGIBILITY:
Inclusion Criteria:

1. The first acute anterior myocardial infarction ( AMI ) within 12 hours ( or more than 12 hours but the ischemic symptoms continue ).
2. Age 18-75 years old, gender unlimited
3. Patients with acute anterior myocardial infarction undergoing emergency PCI within the effective time window
4. Successful reflow after interventional therapy ( TIMI = 3 ).
5. To understand and sign the informed consent.

Exclusion Criteria：

1. Patients with a history of coronary artery bypass grafting
2. Patients with cardiogenic shock
3. Patients with systolic blood pressure ( SBP ) ≤ 90 mmHg after treatment with vasopressors
4. Patients with mechanical complications ( ventricular septal perforation, mitral chordae rupture )
5. Patients with suspected aortic dissection
6. Patients with severe liver and kidney dysfunction
7. Allergic or intolerant to rhBNP.
8. Patients with chronic renal insufficiency requiring long-term dialysis
9. Patients using diuretics during the screening period
10. Pregnant / lactating women
11. Heart diseases that are not suitable for vasodilators, such as severe valve stenosis, restrictive cardiomyopathy, restrictive pericarditis, etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are about 18 to 75 years old get the first acute anterior myocardial infarction ( AMI ) within 12 hours ( or more than 12 hours but the ischemic symptoms continue ) and undergo emergency PCI within the effective time window,after which the blood reflows ( TIMI = 3 ).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
ultrasonic cardiogram：left ventricle ejection fraction (LVEF) | from baseline to 6 months
  LVEF refers to the percentage of stroke output to left ventricular end-diastolic
ultrasonic cardiogram：left ventricular end-diastolic volume index (LVEDVI) | from baseline to 6 months
  LVEDVI（ml/m2）=left ventricular end-diastolic volume（ml）/body surface area
ultrasonic cardiogram：left ventricular end-systolic volume index (LVESVI) | from baseline to 6 months
  LVESVI（ml/m2）=left ventricular end-systolic volume（ml）/body surface area
N terminal pro-B-type natriuretic peptide（NT-proBNP ）decline level | from baseline to 6 months
  NT-proBNP is a protein which is an "ingredient" for making the BNP hormone and a sign of heart failure can be obteined by blood
The level of Cardiac Troponin T(cTnT) | from baseline to 6 months
  The level of Cardiac Troponin T(cTnT) at 6 month

SECONDARY OUTCOMES:
Adverse cardiovascular events | from baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China